CLINICAL TRIAL: NCT05261256
Title: Early Detection of Cardiac Impairments Following Cardiotoxic Anti-cancer Treatment During Childhood and Adolescence - A Feasibility Study
Brief Title: Cardiac Impairments Following Pediatric Cardiotoxic Anti-cancer Treatment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sabine Kesting, Dr. rer. medic., Technical University of Munich
Other Study IDs: German Heart Foundation
Record Dates: First submitted 2021-12-14; First posted 2022-03-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; Pediatric Cancer
Keywords: Childhood cancer; Cardiac impairments; Late effects; Early detection; Prevention; Stress echocardiography
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated for pediatric cancer: This group includes children, adolescents and young adults treated for pediatric cancer who received anthracyclines and/or chest radiation during treatment.
  Interventions: Diagnostic Test: Exercise stress echocardiography
- Healthy control subjects: This group includes healthy children, adolescents and young adults without a history of pediatric cancer as age-and gender-matched control subjects.
  Interventions: Diagnostic Test: Exercise stress echocardiography

INTERVENTIONS:
Diagnostic Test: Exercise stress echocardiography — Study participants perform an exercise stress echocardiography on a semi-supine bicycle ergometer using using a continuous incremental bicycle protocol with a work rate increment every 3 minutes according to gender and weight.

SUMMARY:
This study aims at investigating the feasibility of recruitment and application of a method regarding early detection of subclinical changes in cardiac health after completion of acute cancer treatment during childhood and adolescence.

DETAILED DESCRIPTION:
Cardiovascular late effects following treatment for pediatric cancer are problematic. Early detection of subclinical changes is hardly possible using conventional diagnostic methods, but seems to be feasible during physical strain (exercise stress echocardiography).

This feasibility study examines as main objective the recruitment strategy and investigation method in 10-25-year olds in the first and fifth year after the end of acute anti-cancer therapy (n=40 participants with a history of childhood cancer and n=40 control subjects). The heart function is examined by means of exercise stress echocardiography and spiroergometry in comparison with healthy age- and gender-matched control subjects.

Secondary aims are the evaluation of aditional echocardiography markers and levels of physical activity.

ELIGIBILITY:
Inclusion criteria for all participants:

* Aged between 10 and 25 years
* Body height of ≥1,40m (required for performing the examination on the semi supine bicycle ergometer)
* Signed informed assent (minor participant) and consent (legal guardian and full-aged participant)

Additional inclusion criteria for participants following cancer treatment:

* Completion of acute cancer treatment with anthracyclines and/or chest radiation
* End of treatment 12 months and five years ago (± three months)
* Medical approval for study participation

Additional inclusion criteria for healthy control subjects:

- Appropriate as matched pair with respect to age and gender

Exclusion Criteria:

* Known cardiovascular diseases (incoherent with cardiotoxic treatment)
* Inability to follow study instructions (e.g., mental retardation, language)
* Acute orthopedic injury (e.g., bone fracture) or orthopedic impairments that preclude examination on a bicycle ergometer (e.g., instable prosthetic device)

All participants receive a basic physical and cardiological examination at rest as part of the study protocol to ensure capability before performing the exercise stress echocardiography.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants with a history of pediatric cancer will be recruited during appointments in follow-up care at two departments for pediatric cancer in Munich.
  Healthy peers will be recruited within social environment of participants with a history of cancer (siblings, close friends) and within schools and sport clubs.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Criteria 1 - Recruitment Rate | Throughout study completion, an average of 2 years
  The number of children, adolescents and young adults with a history of pediatric cancer who agree to participate compared to the total number approached for this study.
Feasibility Criteria 2 - Acceptance | Throughout study completion, an average of 2 years
  Number of finished and discontinued exercise stress echocardiographies.
Feasibility Criteria 3 - Data Quality | Throughout study completion, an average of 2 years
  Number of evaluable examination data.
Feasibility Criteria 4 - Practicability | Throughout study completion, an average of 2 years
  Difference between scheduled and required time frame for the single examination.
Feasibility Criteria 5 - Participants' Feedback | Throughout study completion, an average of 2 years
  Feedback questionnaire with multiple choice options and free text answers.

SECONDARY OUTCOMES:
Reference Values of Healthy Peers | Throughout study completion, an average of 2 years
  Assessment of reference values from age- and gender-matched healthy peers (matched pairs).
Analysis of Echocardiography Marker 1 | During the procedure
  Deformation Parameters in % (global longitudinal strain and circumferencial strain)
Analysis of Echocardiography Marker 2 | During the procedure
  Ejection Fraction (EF) in %
Analysis of Echocardiography Marker 3 | During the procedure
  M-Mode Parameter
Analysis of Echocardiography Marker 4 | During the procedure
  Tricuspid Annular Plane Systolic Excursion (TAPSE) in millimeter
Analysis of Echocardiography Marker 5 | During the procedure
  Left ventricle end diastolic volume (LVEDV) in ml/m²
Cardiorespiratory Fitness | During the procedure
  Submaximal oxygen uptake VO2peak (ml/kg/min)
Physical Activity Level post-therapy | During the procedure
  For participants with a history of pediatric cancer: Physical activity questionnaire ActiOn post-therapy for the assessment of the amount of moderate-to-vigorous physical activity.
Physical Activity Level in Healthy Control Subjects | During the procedure
  For healthy control subjects: Physical activity questionnaire from the KiGGS study (German Health Interview and Examination Survey for Children and Adolescents).

CONTACTS AND LOCATIONS:
Overall Officials: Renate Oberhoffer-Fritz, Prof. Dr. med., Study Chair — Institute of Preventive Pediatrics, Department of Sport and Health Sciences, TUM
Locations (1):
- Institute of Preventive Pediatrics, Department of Sport and Health Sciences, Technical University of Munich, Germany, Munich, Germany

IPD SHARING:
Plan to Share IPD: No